CLINICAL TRIAL: NCT05367557
Title: Laparoscopic Surgery: Comparison of Intraoperative Hemodynamic Parameters and Arterial-blood Gas Changes at Two Different Pneumoperitoneal Pressure Values
Brief Title: Comparison of Intraoperative Hemodynamic Parameters and Arterial-blood Gas Changes at Two Different Pneumoperitoneal Pressure Values
Status: Completed | Type: Observational
Sponsor: Eva Intagliata (Other)
Responsible Party: Sponsor-Investigator, Eva Intagliata, researcher, University of Catania
Organization: University of Catania (Other)
Other Study IDs: UCatania000
Record Dates: First submitted 2022-04-14; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Pneumoperitoneum
Keywords: Blood gas analysis alterations; hemodynamic alterations
MeSH Terms: conditions — Pneumoperitoneum | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: pneumoperitoneum pressure of 12 mmHg
  Interventions: Procedure: laparoscopic cholecystectomy
- Group B: pneumoperitoneum pressure of 8 mmHg
  Interventions: Procedure: laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: laparoscopic cholecystectomy — removal of the gallbladder by laparoscopy at pneumoperitoneum pressure setting of 12 or 8 mmHg

SUMMARY:
Clinic and metabolic consequences of pneumoperitoneum, achieved by insufflation of gas carbon dioxide, are still debated. Cardiovascular system suffering due to the compression of intra-abdominal venous structures can cause life-threatening complications. Increased partial pressure of carbon dioxide induces metabolic acidosis with further vascular suffering. Pneumoperitoneum reduces the pulmonary exchange volumes and bring renal suffering.

Methods. The aim of this study is to evaluate the alterations in hemodynamic and hemogasanalysis parameters during the laparoscopic surgery at different pressure settings of pneumoperitoneum in order to assess the best pressure value.

We evaluated and compared intraoperative hemodynamic and hemogasanalytic alterations in two groups of patients respectively subdue to laparoscopic cholecystectomy at a pneumoperitoneum pressure of 12 mmHg (group A) and at a pressure of 8 mmHg (group B).

DETAILED DESCRIPTION:
We evaluated intraoperative hemodynamic and hemogasanalytic alterations in two groups of randomized patients respectively operated at a pneumoperitoneum pressure of 12 mmHg (group A) and at a pressure of 8 mmHg (group B) to highlight any significant alterations.

The clinical sample used in the study is composed by patients aged between 15 and 85 years affected by cholelithiasis and treated with laparoscopic cholecystectomy in the period between July 2019 and February 2020.

20 patients, 9 men and 11 women, were enrolled. Group A included 10 patients, 5 men and 5 women, with an average age of 47.9 years. Group B included 10 patients, 4 men and 6 women, with an average age of 50.7 years.

The parameters evaluated were: heart rate (HR), average arterial blood pressure (BP), respiratory frequency (RF), oxygen saturation (SaO2), hemogasanalysis (PaO2, PaCO2, pH and HCO3-).

The measurements were made at four stages: before the induction of anesthesia, after the anesthesia induction but before incision, 30 minutes after the pneumoperitoneum induction, 5 minutes after the pneumoperitoneum releasing.

The hemodynamic parameters (HR, RF, BP, SaO2) were extrapolated from the multiparameter monitor for each evaluation. The hemogasanalytic values (PaO2, PaCO2, pH and HCO3) were evaluated by the radial arterial sampling. The average and standard deviation were calculated for the quantitative data normally distributed. For the comparison of the quantitative data, the t-student test was used. A value of p ≤ 0,05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria: cholelithiasis -

Exclusion Criteria: immunodeficiency disorders, chronic use of corticosteroids, non-compensated diabetes mellitus, major morbidity with a life expectancy of less than 30 days, significant anemia (hemoglobin < 7 gr/Dl or hematocrit < 21%), coagulopathies, ascites, chronic pain treatment, severe comorbidities

-

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients aged between 15 and 85 years affected by symptomatic cholelithiasis and treated with laparoscopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
hearth rate | before the induction of anesthesia
  hearth rate variations
hearth rate | after the anesthesia induction but before incision
  hearth rate variations
hearth rate | 30 minutes after the pneumoperitoneum induction
  hearth rate variations
hearth rate | 5 minutes after the pneumoperitoneum releasing
  hearth rate variations
arterial blood pressure | before the induction of anesthesia
  average arterial blood pressure variations
arterial blood pressure | after the anesthesia induction but before incision
  average arterial blood pressure variations
arterial blood pressure | 30 minutes after the pneumoperitoneum induction
  average arterial blood pressure variations
arterial blood pressure | 5 minutes after the pneumoperitoneum releasing
  average arterial blood pressure variations
respiratory frequency | before the induction of anesthesia
  respiratory frequency variations
respiratory frequency | after the anesthesia induction but before incision
  respiratory frequency variations
respiratory frequency | 30 minutes after the pneumoperitoneum induction
  respiratory frequency variations
respiratory frequency | 5 minutes after the pneumoperitoneum releasing
  respiratory frequency variations
oxygen saturation | before the induction of anesthesia
  oxygen saturation variations
oxygen saturation | after the anesthesia induction but before incision
  oxygen saturation variations
oxygen saturation | 30 minutes after the pneumoperitoneum induction
  oxygen saturation variations
oxygen saturation | 5 minutes after the pneumoperitoneum releasing
  oxygen saturation variations
blood gas analysis | before the induction of anesthesia
  blood gas analysis variations
blood gas analysis | after the anesthesia induction but before incision
  blood gas analysis variations
blood gas analysis | 30 minutes after the pneumoperitoneum induction
  blood gas analysis variations
blood gas analysis | 5 minutes after the pneumoperitoneum releasing
  blood gas analysis variations

CONTACTS AND LOCATIONS:
Locations (1):
- Eva Intagliata, Catania, Italy

IPD SHARING:
Plan to Share IPD: No